CLINICAL TRIAL: NCT05604274
Title: Longitudinal Monitoring of Stool Characteristics
Status: Completed | Type: Observational
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: BAJAJ033
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbiome analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls
  Interventions: Other: App to monitor stool consistency and symptoms
- Patients with cirrhosis on lactulose
  Interventions: Other: App to monitor stool consistency and symptoms
- Patients with cirrhosis on rifaximin
  Interventions: Other: App to monitor stool consistency and symptoms

INTERVENTIONS:
Other: App to monitor stool consistency and symptoms — App to monitor stool consistency and symptoms

SUMMARY:
In patients with cirrhosis and healthy controls to determine the utility of an App to classify BSS compared to assessment made by the patients themselves using the BSS and correlate these with other stool characteristics and gut microbiota.

DETAILED DESCRIPTION:
In patients with cirrhosis and healthy controls to determine the utility of an App to classify BSS compared to assessment made by the patients themselves using the BSS and correlate these with other stool characteristics and gut microbiota.

Patients with cirrhosis are often treated with lactulose, that needs monitoring of bowel movement numbers and is overall not acceptable to a majority of patients. The estimation of this number is not completely accurate and varies day by day. In addition, recent work has shown that consistency of the stools with the Bristol Stool Scale (BSS) may be another important metric to determine who will respond well to lactulose versus not.

In addition to the issue of remembering exact details of bowel movement frequency, it is often hard for patients, especially with HE, to remember details of their daily function. Additionally, insight into the impact of the disease. Traditionally, patients assess stool form and consistency using the Bristol stool score and chart, which classifies stool into one of seven types. A challenge with this is that the assessment is subjective and may vary from patient to patient. This is seen in patients without cognitive dysfunction such as those with irritable bowel syndrome (IBS). Therefore, it is likely that patients with cirrhosis, who often have cognitive dysfunction, could be worse in estimating stool consistency. In addition, microbiome structure and function, which is often dependent on stool consistency may be measured differently based on personal vs app-generated BSS values.

Thus, method to better estimate stool characteristics, which could better inform patient management through telemedicine is needed. Aim: Monitor patients using a mobile health application designed for monitoring and assessing patients with digestive diseases.

ELIGIBILITY:
Inclusion Criteria:

* For cirrhosis subjects must meet all of the following inclusion criteria to be eligible:

  1. Male and female subjects aged ≥ 18 years.
  2. Cirrhosis
  3. Able and willing to voluntarily complete the informed consent process
  4. Familiar with smartphone technology
  5. Available for and agree to all study procedures, including taking the pictures of the stool and collection of stool

For controls :

1. Male and female subjects aged ≥ 18 years.
2. Absence of chronic diseases requiring prescription medications
3. Able and willing to voluntarily complete the informed consent process
4. Familiar with smartphone technology
5. Available for and agree to all study procedures, including taking the pictures of the stool and collection of stool for microbiome analysis

Exclusion Criteria:

Subjects with cirrhosis meeting any of the following criteria are not eligible for study enrollment:

1. Unclear diagnosis of cirrhosis
2. History of liver transplant
3. For those on lactulose, they need to be on it for at least 2 weeks
4. Unfamiliar with smartphones
5. Apart from chronic liver disease, any acute or chronic medical, surgical, psychiatric, or social condition including history of cerebrovascular disease (stroke, transient ischemic attack) or dementia, that may increase the subject risk associated with study participation, compromise adherence to study procedures and requirements, confound interpretation of the results, and, in the judgment of the investigator, make the subject inappropriate for enrollment.

For healthy controls

1. Any chronic disease requiring prescription medications
2. Unfamiliar with smartphones

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified through word of mouth or through clinic evaluations and approached to participate in this study. Their medications, clinical and medical history will be recorded to determine eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
App use comfort measured by survey | 2 weeks
  A survey designed to assess acceptability of this App at baseline and at 2 weeks; higher score=good

SECONDARY OUTCOMES:
Quality of life using Sickness Impact Profile | 2 weeks
  we will test association of the stool characteristics with quality of life; higher=good
Cognitive testing using PHES | 2 weeks
  we will test association of the stool characteristics with PHES values; higher=good
Alpha diversity using Shannon index of microbiome | 2 weeks
  we will test association of the stool characteristics with microbial characteristics
Bristol stool scale by subjects | 2 weeks
  we will test association of the stool characteristics gauged through the App versus the Bristol stool scale by subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fagan A, Gallagher ML, Mousel T, Davis BC, Fuchs M, Puri P, Anstey J, Tiede D, Simonetto DA, Kraus A, Bajaj JS. Artificial Intelligence Evaluation of Stool Quality Guides Management of Hepatic Encephalopathy Using a Smartphone App. Am J Gastroenterol. 2024 May 1;119(5):977-981. doi: 10.14309/ajg.0000000000002646. Epub 2023 Dec 28. PMID 38153339

DOCUMENTS (1):
  • Informed Consent Form (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT05604274/ICF_000.pdf